CLINICAL TRIAL: NCT07359703
Title: A Prospective Study to Evaluate the Outcome of the Aurora Test Used With Blastocyst Transfer in an ICSI Cycle
Brief Title: A Prospective Study to Evaluate the Outcome of the Aurora Test Used With Blastocyst Transfer in an ICSI Cycle (Aurora-Blasto)
Acronym: Aurora-Blasto
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Fertiga, Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ONZ-2024-0423; 12947 (Other: UZ Ghent Ethical committee)
Record Dates: First submitted 2025-09-08; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: ART

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Informative subjects (i.e., prospective data): patients undergoing ICSI treatment (Experimental): The Department of Reproductive Medicine is initiating a clinical study to investigate a new test called the Aurora test. This test uses cells that surround the woman's egg. These cells are normally not usable, as they are separated from the egg and discarded. However, for the Aurora test, these cells are not discarded but instead used for analysis.
  Patients undergo standard of care treatment in addition to the Aurora-test. The Aurora test is designed to score the embryos obtained. This score indicates which embryo has the highest chance of leading to a pregnancy. After the embryologist selects the embryos for transfer, the Aurora test will determine the order of transfer. The tested embryos will receive an Aurora test score from high to low, with the highest-scoring embryos being transferred first. As a result, the Aurora test may help people become pregnant more quickly.
  Interventions: Other: Aurora-Blasto

INTERVENTIONS:
Other: Aurora-Blasto — The Department of Reproductive Medicine is initiating a clinical study to investigate a new test called the Aurora test. This test uses cells that surround the woman's egg. These cells are normally not usable, as they are separated from the egg and discarded. However, for the Aurora test, these cells are not discarded but instead used for analysis. Patients undergo standard of care treatment in addition to the Aurora-test. The Aurora test is designed to score the embryos obtained. This score indicates which embryo has the highest chance of leading to a pregnancy. After the embryologist selects the embryos for transfer, the Aurora test will determine the order of transfer. The tested embryos will receive an Aurora test score from high to low, with the highest-scoring embryos being transferred first. As a result, the Aurora test may help people become pregnant more quickly.

SUMMARY:
In current treatments for In Vitro Fertilization (IVF) and Intracytoplasmic Sperm Injection (ICSI), the creation of multiple embryos is a common practice. The decision to transfer an embryo is traditionally based on the morphological assessment by an embryologist, which, due to its nature, must be considered subjective. In certain regions, invasive embryo biopsy techniques, such as Preimplantation Genetic Testing for Aneuploidy (PGT-A), are used to detect chromosomal abnormalities and support decision-making regarding embryo transfer. However, there is a medical need to improve the outcomes of IVF/ICSI cycles through non-invasive and objective methods.

As an academic center, our goal is to investigate promising innovative methods that, if successful, can be integrated into standard care. The aim of the Aurora blastocyst study is to evaluate the effectiveness of the Aurora test in selecting five-day-old embryos for fresh or frozen embryo transfer. Additionally, the study assesses whether the use of the Aurora test results in an increase in clinical pregnancy rates and live birth rates.

The Aurora test is a non-invasive test for evaluating oocyte competence and subsequently the embryo obtained in an ICSI cycle (In Vitro Fertilization). This test is performed on cumulus cells (CC) surrounding the oocyte and uses mRNA expression profiles to evaluate the developmental potential of the oocytes. The test has been developed and validated for patients stimulated with human menopausal gonadotropins (HP-hMG), an ovulatory dose of hCG, and a single embryo transfer on day 3. The test will be performed by Fertiga nv, upon receiving patients cumulus cells.

At our center, based on earlier research, the standard care involves a single embryo transfer on day 5. In this study, embryo selection based on morphology is compared with embryo selection based on morphology and the Aurora test. Finally, this study aims to evaluate the impact of the Aurora test score on the embryologist's selection decision for transferring a five-day-old embryo for single embryo transfer, by assessing parameters such as pregnancy rates and live birth rates.

DETAILED DESCRIPTION:
The only additional procedure involves analyzing waste material i.e. cumulus cells by Fertiga nv. RNA is extracted from the cumulus cells and analyzed using qRT-PCR. Cumulus cells iare then assigned to a score based on its RNA levels. This score, known as the Aurora test score, indicates the pregnancy potential of the associated oocyte. Using this evaluation, the embryologist will select the best embryo candidates for transfer. The embryo with the highest Aurora test score from this group will be transferred. If there is no live birth and the trial has not been concluded, the patient may consider frozen/thawed embryo transfer cycles. These consecutive frozen/thawed embryo transfer cycles will also be based on the Aurora test score.

The two experimental arms (i.e. fresh SET and frozen/thawed SET) will each include approximately 140 informative patients prospectively recruited for the study undergoing ICSI, with a day 5 blastocyst transfer chosen by embryo morphology and Aurora Test. Taking into account a dropout rate of 40%, 234 patients will be required in each experimental arm. All patients in the experimental arm need to fulfil the inclusion and exclusion criteria as detailed in the protocol. The patients signing the informed consent form (ICF) will have their Cumulus Oocyte complex (COC) numbered at oocyte pick-up (OPU), tracked individually, cumulus cells will be individually denuded and then be snap-frozen and analysed for mRNA expression using oocyte quality predictive genes and two control genes. The RNA expression analysis will be done at Fertiga's Molecular Laboratory. The lab technician/embryologist will track the individual embryos during their growth as usual and classify the embryos based on their routine morphological quality parameters. From the embryos considered for transfer i.e. based on the morphology grading, the one with the highest Aurora Test ranking will be selected for single blastocyst transfer.

The study will use two matched historical control groups, each containing 280 patients, resulting in 560 control patients treated within the last 4 years at the Department of Reproductive Medicine of Ghent University Hospital preceding the initiation of the current study (retrospective study cohort). All control patients need to fulfil all the inclusion and exclusion criteria. These control patients will be matched controls where each patient undergoing the Aurora Test will be matched with two patients that had a single embryo transfer based only on morphological grading features. The controls will be matched for stimulation protocol, transfer regime (fresh or frozen/thawed), ovulation trigger (hCG/dual trigger/GnRH agonist), age category (<31, 31-35, >35) and for number of good/top quality D5 embryos (2/ 3-4 / 5-6 / >6).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ICSI treatment, with maximum 40 years of age at time of signing the ICF
2. Patients stimulated with GnRH antagonist/HP-hMG or GnRH antagonist/recFSH, scheduled for fresh SET Day 5 with hCG or dual trigger (hCG + GnRH agonist) or Patients stimulated with GnRH antagonist/HP-hMG or GnRH antagonist/recFSH, scheduled for delayed transfer of frozen/thawed SET Day 5 after a GnRH agonist trigger, hCG or dual trigger (hCG + GnRH agonist).
3. Patients undergoing a first, second, third or fourth ICSI cycle
4. Women with body mass index (BMI) higher than 17 and lower than 35
5. Women with regular cycles (between 24 and 35 days)
6. Non-and mild-smokers (<10 cigarettes/day)
7. AMH 1,1 ng/ml (Bologna criteria), excluding poor responders according to Bologna criteria
8. Patients with fresh ejaculated semen or frozen donor semen

Exclusion Criteria:

1. Patients with less than 8 follicles (≥12mm) on the day of their last echo visit before OPU.
2. Women with history of poor oocyte maturation in a previous cycle (< 50% MII)
3. Women with Severe Endometriosis (≥ III AFS classification) (in the ovaries and if not surgically treated)
4. Patients scheduled for PGD (preimplantation genetic diagnosis of monogenic/single gene defects) and PGT-A (preimplantation genetic testing on aneuploidy)
5. Couples where the partner has an extremely low sperm count e.g.: severe oligo-astheno-teratozoospermia (OAT) with sperm count below 100.000/ml or TESE.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1028 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Blastocyst selection | At Day 5 of the embryodevelopment, which is 5 days after Oocyte retrieval and ICSI procedure (D0). The Oocyte retrieval occurs after the ICF has been signed.
  The primary objective of the study is to demonstrate a significant difference between selection of blastocysts solely based on morphology versus selection of the blastocyst guided by a combination of morphology and the Aurora Test ranking. We assume that the difference between the two ranking methods will be observed in at least 30% of the patients.

SECONDARY OUTCOMES:
Clinical Pregnancy Rate | From enrollment to pregnancy confirmed by ultrasound or clinical evidence of at least one fetus with a detectable heartbeat between weeks 6 and 8
  The secondary objective is to evaluate the increase of Clinical Pregnancy Rate in the experimental arm where transfer of a single blastocyst at Day 5 is based on the Aurora Test score in combination with morphological selection compared to morphological selection alone in the historical matched control arm .

OTHER OUTCOMES:
Ongoing Pregnancy Rate (OPR) in the experimental arms versus historical control arm | From enrollment to pregnancy confirmed by ultrasound or clinical evidence of at least one gestational sacs with fetal heart beat between weeks 10 and 12.
  Ongoing Pregnancy Rate (OPR) in the experimental arms versus historical control arm for a Single Embryo Transfer (SET) of Day 5 embryos (while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).
Increase LBR in the experimental arms vs. the historical control arm | From enrollment (i.e. study start), which is directly followed by Oocyte retrieval (D0) to childbirth, approximately 9 months after the transfer of a Day 5 embryo.
  Increase of the Live Birth Rate (LBR) in the experimental arms versus the historical control arm for a SET of Day 5 embryos (while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).
CPR, OPR and LBR | From enrollment (i.e. study start), which is directly followed by Oocyte retrieval (D0) to childbirth, approximately 9 months after the transfer of a Day 5 embryo.
  Clinical Pregnancy Rate (CPR), OPR and LBR with respect to number of oocytes at pick-up, number of transferable embryos at Day 3, number of blastocysts at Day 5 (while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).
CPR, OPR and LBR in different age groups | From enrollment (i.e. study start), which is directly followed by Oocyte retrieval (D0) to childbirth, approximately 9 months after the transfer of a Day 5 embryo.
  CPR, OPR and LBR in age group 22-34 years, in age group 35-37 years, and in age group 38-40 years (while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).
TTP and CPR | From enrollment (i.e. study start), which is directly followed by Oocyte retrieval (D0) to childbirth, approximately 9 months after the transfer of a Day 5 embryo.
  Time to pregnancy and cumulative pregnancy rates (i.e. Clinical Pregnancy, Ongoing Pregnancy, Live Birth; while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).
Aurora Test VS iDA/KID score ranking | From enrollment (i.e. study start), which is directly followed by Oocyte retrieval (D0) to childbirth, approximately 9 months after the transfer of a Day 5 embryo.
  Compare the Aurora Test ranking with the iDA /KID Score ranking of the transferable embryos, for the patients with embryos grown in the Embryoscope (while taking into account the patient stimulation (HP-hMG or rFSH ) and ovulation trigger).

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium